CLINICAL TRIAL: NCT03975088
Title: Sub-macular Injection of Ranibizumab as a New Surgical Treatment for Refractory Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alexandria (Other)
Responsible Party: Principal Investigator, Mahmoud Abouhussein, Assistant professor, University of Alexandria
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 31185
Record Dates: First submitted 2019-06-02; First posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persistent Diabetic macular edema (Other): Authors defined refractory DME as eyes with persistent DME despite receiving at least 6 monthly Ranibizumab injections of anti VEGF, and then switched to Aflibercept, receiving at least three monthly injections.
  Interventions: Procedure: Sub-macular injection of Ranibizumab

INTERVENTIONS:
Procedure: Sub-macular injection of Ranibizumab — In this study, authors describe a new surgical technique for the treatment of refractory non tractional DME. The technique consists of vitrectomy with ILM peeling with subretinal injection of Ranibizumab.

SUMMARY:
The best treatment strategy for refractory DME is not known, options include switching between anti-VEGF agents, corticosteroids, and vitrectomy. In this study, authors describe a new surgical technique for the treatment of refractory non tractional DME. The technique consists of vitrectomy with ILM peeling with subretinal injection of Ranibizumab.

DETAILED DESCRIPTION:
Purpose: In this study, authors describe a new surgical technique for the treatment of refractory DME. The technique consists of vitrectomy with ILM peeling with subretinal injection of Ranibizumab.

Methods: This is a prospective interventional non-comparative study including patients with refractory DME. Included patients were subjected to the new surgical technique of pars plana vitrectomy with sub-retinal injection of Ranibizumab.

ELIGIBILITY:
Inclusion Criteria:

* refractory diffuse non tractional DME.
* Central retinal thickness (CRT) should exceed 350 µm despite undergoing multiple anti-VEGF therapy.
* Decimal best corrected visual acuity (BCVA) must be ≥0.01 and ≤0.5.

Exclusion Criteria:

* Previous vitrectomy, recent cataract surgery less than 6 months,
* evident RPE atrophy, proliferative diabetic retinopathy, massive foveal hard exudation, foveal traction on OCT,
* glaucoma and one eyed patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The primary endpoint for this study was the change in CMT at the final visit. | at the 6 month follow up visit
  Central macular thickness

IPD SHARING:
Plan to Share IPD: No
proecting patient privacy

REFERENCES:
- [Derived] El-Baha SM, Abdel Hadi AM, Abouhussein MA. Submacular Injection of Ranibizumab as a New Surgical Treatment for Refractory Diabetic Macular Edema. J Ophthalmol. 2019 Oct 21;2019:6274209. doi: 10.1155/2019/6274209. eCollection 2019. PMID 31772766